CLINICAL TRIAL: NCT02064582
Title: Phase 2 Study of Enzalutamide and GnRH Agonist Before, During and After Radiation Therapy in Treatment of Patients With High-risk Localized Prostate Cancer
Brief Title: Enzalutamide and Hormone Therapy Before, During, and After Radiation for High Risk Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Principal Investigator, Kevin Dale Courtney, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 082013-032
Record Dates: First submitted 2014-02-10; First posted 2014-02-17 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-09

CONDITIONS: Prostate Cancer
Keywords: prostate cancer, enzalutamide, radiation, hormone therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Leuprolide; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Enzalutamide, Leuprolide, radiation (Other): Single arm Enzalutamide 160 mg daily for 6 months Leuprolide acetate 22.5mg every 3 months or 45mg every 6 months Radiation therapy as standard of care
  Interventions: Drug: Enzalutamide; Drug: Leuprolide acetate; Radiation: radiation

INTERVENTIONS:
Drug: Enzalutamide — 160mg by mouth each day
  Other Names: Xtandi
Drug: Leuprolide acetate — 22.5 mg intramuscular every 3 months or 45mg intramuscular every 6 months
  Other Names: Lupron
Radiation: radiation — External beam radiation will be delivered as per standard radiation therapy protocol

SUMMARY:
The study is being done to find out whether combining two FDA approved drugs along with radiation therapy for the treatment of high risk localized prostate cancer is safe and well tolerated.

DETAILED DESCRIPTION:
* this pilot study will assess the safety and tolerability of combining enzalutamide with an gonadotropin-releasing hormone agonist (GnRH) and external beam radiation
* Correlative imaging and tissue biopsy analysis will be performed to assess the radiographic response to enzalutamide plus gonadotropin-releasing hormone agonist (GnRH) therapy as well as intratumoral androgen signaling

ELIGIBILITY:
Inclusion Criteria:

* histologically proven adenocarcinoma of the prostate within 6 months of screening
* Eastern Cooperative Oncology Group(ECOG) score 0-2
* adequate organ and and blood marrow function
* must be a candidate for long-term androgen deprivation in combination with external beam radiation for the treatment of high risk prostate cancer
* patient must permit a targeted prostate biopsy at the time of study initiation or at the beginning of radiation treatment
* men who are sexually active with female partners of child-bearing potential mush agree to use adequate contraception

Exclusion Criteria:

* prior treatment with agents known to have endocrine effects on prostate cancer
* treatment with corticosteroids within 4 weeks of enrollment
* treatment with androgens within 6 months of enrollment
* may not be receiving any other investigational agents
* Prostate specific antigen greater than 160ng/dL
* history of malignancy( other than non-melanoma skin cancer) within 5 years
* uncontrolled intercurrent illness
* cardiovascular event within 6 months of enrollment
* seizure or seizure disorder history
* contraindications to MRI- pacemakers, clips, etc

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-06-09 (Actual); Study Completion 2018-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin D Courtney, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Li J, Alyamani M, Zhang A, Chang KH, Berk M, Li Z, Zhu Z, Petro M, Magi-Galluzzi C, Taplin ME, Garcia JA, Courtney K, Klein EA, Sharifi N. Aberrant corticosteroid metabolism in tumor cells enables GR takeover in enzalutamide resistant prostate cancer. Elife. 2017 Feb 13;6:e20183. doi: 10.7554/eLife.20183. PMID 28191869

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 7 met criteria and were enrolled in the trial
Period: Overall Study
Arm/Group | Enzalutamide, Leuprolide, Radiation
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Enzalutamide, Leuprolide, Radiation
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Safety, as Measured by the Number of Patients With at Least One Adverse Event as Assess by NCI Common Terminology Criteria for Adverse Events (CTCAE) vs. 40 When Combining Enzalutamide With a GnRH and External Beam Radiation
Description: Assessment will number of participants who experience adverse events greater than or equal to Grade 3, as defined by NCI Common terminology criteria for adverse events(CTCAE) v4.0
Time Frame: 12 months following initiation of treatment with enzalutamide plus GnRH agonist
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide, Leuprolide, Radiation
Number analyzed (Participants) | 7
Participants | 0

2. Secondary Outcome: Fold Change in Intra-tumoral Androgen Regulated Gene Expression Pre and Post Combination Therapy
Description: Fold change of Intra-tumoral Androgen Regulated Gene Expression (PSA, FKBP5, TMPRSS2, and NDRG1) will be measure at 12 months post therapy.
Time Frame: 12 months
Measure: Median (Full Range); unit: Fold change
Arm/Group | Enzalutamide, Leuprolide, Radiation
Number analyzed (Participants) | 7
Fold change
  Fold change in PSA | 0.54 [0.16 to 21]
  Fold change in FKBP5 | 2.2 [0.72 to 22.15]
  Fold change in TMPRSS2 | 0.65 [0.17 to 3.3]
  Fold change in NDRG1 | 0.36 [0 to 7.53]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of consent and ended 30 days post medication, an average of one year
Arm/Group | Enzalutamide, Leuprolide, Radiation
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide, Leuprolide, Radiation (N=7)
Abdominal pain / bloating (Gastrointestinal disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Aneurysm internal iliac artery (Vascular disorders) | 1 (1)
Anxiety / depression (Psychiatric disorders) | 2 (2)
Lower extremity edema (Musculoskeletal and connective tissue disorders) | 3 (3)
Blurred vision (Eye disorders) | 3 (3)
constipation (Gastrointestinal disorders) | 4 (4)
fatigue (General disorders) | 6 (6)
hot flashes / night sweats (General disorders) | 7 (8)
Diarrhea / loose stools (Gastrointestinal disorders) | 4 (7)
Heartburn (Gastrointestinal disorders) | 2 (2)
Dizziness (General disorders) | 3 (3)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Joint pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Bone metastasis (General disorders) | 1 (1)
Bruit of left carotid artery (Cardiac disorders) | 1 (1)
Cataract, both eyes (Eye disorders) | 1 (1)
Change in mole on neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Clammy skin, oiliness, filminess skin/teeth (Skin and subcutaneous tissue disorders) | 1 (2)
Chest pain (General disorders) | 1 (1)
Lower back pain (General disorders) | 1 (1)
Color perception changes (Eye disorders) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Neuropathy (Skin and subcutaneous tissue disorders) | 5 (5)
Decrease in energy (General disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Decreased night vision (Eye disorders) | 1 (1)
Emotional depression/insomina (Psychiatric disorders) | 1 (1)
Erectile dysfunction (General disorders) | 1 (1)
Fall (General disorders) | 1 (1)
Folliculitis (General disorders) | 1 (1)
Frontal headaches (General disorders) | 1 (1)
Hearing loss (Ear and labyrinth disorders) | 1 (1)
Hematochezia (Gastrointestinal disorders) | 2 (2)
Noctoria (Renal and urinary disorders) | 3 (4)
burning on urination (Renal and urinary disorders) | 1 (1)
Nausea (General disorders) | 2 (2)
Hoarseness/ fullness in throat (General disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Weight gain (General disorders) | 2 (2)
Hot flashes with sweating/night sweats (General disorders) | 1 (1)
Hyperglycemia (Endocrine disorders) | 2 (2)
Vivid dreams (General disorders) | 1 (1)
Increased hunger (General disorders) | 1 (1)
Urethral pain/ dysuria (Renal and urinary disorders) | 3 (3)
Urinary dribbling (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 4 (4)
Lightheadedness (General disorders) | 2 (2)
Lower back pain (General disorders) | 2 (2)
Loss of smell (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bone / joint pain (Musculoskeletal and connective tissue disorders) | 7 (7)
Left pectoralis skin lesion bx squamous cell (Skin and subcutaneous tissue disorders) | 1 (1)
Transaminitis (Hepatobiliary disorders) | 3 (3)
Morning Stiffness/ arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Internal tension (General disorders) | 1 (1)
Memory loss (General disorders) | 1 (1)
Muscle pull left wrist (Musculoskeletal and connective tissue disorders) | 1 (1)
Adenopathy (Blood and lymphatic system disorders) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pelvic pain/prostate/ inguinal (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Poor appetite (Metabolism and nutrition disorders) | 1 (1)
Radiation proctitis (Surgical and medical procedures) | 1 (1)
Rectal burning / irritation (General disorders) | 2 (2)
Recurrence of claudication in setting of PVD (General disorders) | 1 (1)
Right breast tenderness and swelling (General disorders) | 1 (1)
Short term memory impairment (General disorders) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 2 (2)
Ringing in ears (Endocrine disorders) | 1 (1)
Seasonal Allergies (General disorders) | 1 (1)
Spontaneous passage of kidney stone (General disorders) | 1 (1)
Stress Incontinence (General disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Vomiting (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-12-29): https://cdn.clinicaltrials.gov/large-docs/82/NCT02064582/Prot_SAP_000.pdf
  • Informed Consent Form (2016-08-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT02064582/ICF_001.pdf